CLINICAL TRIAL: NCT07143656
Title: Natural History and Biomarker Correlation Study in Amyotrophic Lateral Sclerosis: A Multicenter Retrospective Observational Registry
Brief Title: Amyotrophic Lateral Sclerosis: A Multicenter Retrospective Observational Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Biocells Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Bio120003
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Amyotrophic Lateral Sclerosis &Amp; Other Neuromuscular Disorders
Keywords: Amyotrophic Lateral Sclerosis; MSC; biomedicine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Imaging and Clinical Reports — Inclusion of existing imaging data (MRI, EMG reports) and standard clinical documentation, where available.

SUMMARY:
This retrospective observational study will analyze de-identified clinical data from patients with amyotrophic lateral sclerosis (ALS) collected at multiple centers over 7 years. The primary objective is to describe disease progression using the ALS Functional Rating Scale-Revised (ALSFRS-R). Secondary objectives include evaluating survival, ventilatory decline, and correlations between available biomarkers (e.g., neurofilament light chain, cytokines) and disease trajectory. No new interventions or patient contact will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of amyotrophic lateral sclerosis (ALS) or motor neuron disease confirmed.
2. Age ≥18 years.
3. Availability of at least one ALS Functional Rating Scale-Revised (ALSFRS-R) score.
4. Availability of longitudinal follow-up data.

Exclusion Criteria:

1. Patients with alternative diagnoses that mimic ALS (e.g., multifocal motor neuropathy, cervical myelopathy, myasthenia gravis).
2. Absence of medical records

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged ≥18 with ALS
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2028-08-13 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in ALS Functional Rating Scale-Revised (ALSFRS-R) scores | 2 yearss after the first administration
  Unit: points per month

CONTACTS AND LOCATIONS:
Locations (1):
- Biocells Medical, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No